CLINICAL TRIAL: NCT03417063
Title: Intracranial Artery Stenosis Magnetic Resonance Imaging: Aetiology and Progression (ICASMAP)
Brief Title: Intracranial Artery Stenosis Magnetic Resonance Imaging: Aetiology and Progression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Tiantan Hospital (Other); Beijing Hospital (Other Government); 309th Hospital of Chinese People's Liberation Army (Other); Navy General Hospital, Beijing (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); Beijing Huairou Hospital (Other); Beijing Pinggu District Hospital (Other); Beijing Shuyi Hospital (Other); Tianjin First Central Hospital (Other); Tianjin 4th Centre Hospital (Unknown); Tianjin Union Medical Center (Other); Hebei Medical University Third Hospital (Other); Affiliated Hospital of Chengde Medical University (Other); Tangshan Gongren Hospital (Other); The First Affiliated Hospital of Hebei North University (Other); Cangzhou People's Hospital (Other); Harrison International Peace Hospital (Other)
Responsible Party: Principal Investigator, Xihai Zhao, Professor, Tsinghua University
Other Study IDs: D171100003017003
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Intracranial Artery Stenosis
Keywords: Intracranial artery; Atherosclerosis; Intracranial artery stenosis; High-Resolution Magnetic Resonance
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke has become the leading cause of death in China. It has been shown that intracranial artery stenosis (ICAS) plays a key role in Chinese stroke patients. Although most of stenotic diseases in intracranial arteries are atherosclerotic, a substantial number of other vascular diseases, such as dissection, arteritis, moyamoya disease, and reversible cerebral vasoconstriction syndrome (RCVS), can also lead to intracranial artery luminal narrowing. It is challenging to differentiate the etiologies of ICAS relying on measuring luminal narrowing by angiographical approaches. In addition, the progression of intracranial atherosclerotic disease (ICAD) has been demonstrated to be highly associated with the risk of ischemic cerebrovascular events. However, the influence factors for ICAD progression remains unclear.

High-resolution magnetic resonance imaging (HR-MRI) has been widely used to assess ICAS diseases. The different etiologies of ICAS are differentiable by MR-MRI according to the features of location, shape, signal pattern, remodeling, and contrast enhancement. Investigators have proved that HR-MRI is a reproducible technique that may be reliably utilized to monitor the changes of ICAD during natural follow-up or medical treatment.

The ICASMAP (Intracranial Artery Stenosis MR Imaging: Aetiology and Progression) is a prospective, cross-sectional, observational, and multicenter study. The objectives of ICASMAP are to determine: 1) the spectrum of etiology of ICAS in stroke patients; and 2) the influence factors for progression of ICAD. A total of 300 patients with symptomatic stenotic disease in intracranial arteries (stenosis range: 30%-99%) will be recruited within two weeks after symptom onset from 18 different hospitals across Beijing-Tianjin-Hebei region in China within 1 year. All the patients will undergo HR-MRI for intracranial arteries at baseline, one-year, and two-years. The clinical risk factors will be collected and blood draw will be conducted. The ICASMAP study may help to improve the precise diagnosis and intervention of ICAS and stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent transient ischemic attack or ischemic stoke within two weeks after symptom onset and intracranial artery stenosis (30%-99%) at least in intracranial internal carotid artery,basilar artery, M1 segment of middle cerebral artery , A1 segment of anterior cerebral artery, or P1 segment of posterior cerebral artery determined by computed tomography angiography or magnetic resonance (MR) angiography.

Exclusion Criteria:

* Patients with specific carotid artery atherosclerotic plaques
* Patients with evidence of may causing cardiac thrombosis disease
* Patients with claustrophobia
* Patients with contraindications to MR imaging
* Patients with heart or respiratory failure
* Patients with renal insufficiency (serum creatinine >133umol/L)
* Patients with serious disturbance of consciousness
* Patients with brain tumors
* Patients with cerebral hemorrhage
* Pregnant woman or plan to pregnant within recent 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, we plan to recruit patients with recent transient ischemic attack or ischemic stoke within two weeks after symptom onset and intracranial artery stenosis (30%-99%) at least in intracranial internal carotid artery,basilar artery, M1 segment of middle cerebral artery, A1 segment of anterior cerebral artery, or P1 segment of posterior cerebral artery determined by computed tomography angiography or magnetic resonance angiography. The patients will be recruited from 18 hospitals in Beijing-Tianjin-Hebei area of China.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-14 (Actual); Primary Completion 2021-03-25 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
Progression of plaque burden | 24 months
  Maximum wall thickness

SECONDARY OUTCOMES:
Progression of luminal stenosis | 24 months
  Mild (<50%), moderate (50-70%), severe (70-99%), and occlusion
Progression of plaque components | 24 months
  Presence of intraplaque hemorrhage
cerebrovascular events | 24 months
  ischemic stroke or transient ischemia attack

CONTACTS AND LOCATIONS:
Overall Officials: Xihai Zhao, MD, PhD, Principal Investigator — Tsinghua University
Locations (1):
- Center for Biomedical Imaging Research, Department of Biomedical Engineering, Tsinghua University, Beijing, China

REFERENCES:
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Ahn SH, Lee J, Kim YJ, Kwon SU, Lee D, Jung SC, Kang DW, Kim JS. Isolated MCA disease in patients without significant atherosclerotic risk factors: a high-resolution magnetic resonance imaging study. Stroke. 2015 Mar;46(3):697-703. doi: 10.1161/STROKEAHA.114.008181. Epub 2015 Jan 27. PMID 25628303
- [Background] Hart RG, Diener HC, Coutts SB, Easton JD, Granger CB, O'Donnell MJ, Sacco RL, Connolly SJ; Cryptogenic Stroke/ESUS International Working Group. Embolic strokes of undetermined source: the case for a new clinical construct. Lancet Neurol. 2014 Apr;13(4):429-38. doi: 10.1016/S1474-4422(13)70310-7. PMID 24646875
- [Background] Wang Y, Xu J, Zhao X, Wang D, Wang C, Liu L, Wang A, Meng X, Li H, Wang Y. Association of hypertension with stroke recurrence depends on ischemic stroke subtype. Stroke. 2013 May;44(5):1232-7. doi: 10.1161/STROKEAHA.111.000302. Epub 2013 Feb 26. PMID 23444308
- [Background] Gorelick PB, Wong KS, Bae HJ, Pandey DK. Large artery intracranial occlusive disease: a large worldwide burden but a relatively neglected frontier. Stroke. 2008 Aug;39(8):2396-9. doi: 10.1161/STROKEAHA.107.505776. Epub 2008 Jun 5. PMID 18535283
- [Background] Choi YJ, Jung SC, Lee DH. Vessel Wall Imaging of the Intracranial and Cervical Carotid Arteries. J Stroke. 2015 Sep;17(3):238-55. doi: 10.5853/jos.2015.17.3.238. Epub 2015 Sep 30. PMID 26437991
- [Background] Mossa-Basha M, Hwang WD, De Havenon A, Hippe D, Balu N, Becker KJ, Tirschwell DT, Hatsukami T, Anzai Y, Yuan C. Multicontrast high-resolution vessel wall magnetic resonance imaging and its value in differentiating intracranial vasculopathic processes. Stroke. 2015 Jun;46(6):1567-73. doi: 10.1161/STROKEAHA.115.009037. Epub 2015 May 7. PMID 25953365
- [Derived] Han Y, Zhang R, Yang D, Li D, Han H, Qiao H, Chen S, Wang Y, Yu M, Hong Y, Wang Z, Zhao X, Liu G. Risk Factors for Asymptomatic and Symptomatic Intracranial Atherosclerosis Determined by Magnetic Resonance Vessel Wall Imaging in Chinese Population: A Case-Control Study. Ther Clin Risk Manag. 2022 Jan 12;18:61-70. doi: 10.2147/TCRM.S335401. eCollection 2022. PMID 35058694